CLINICAL TRIAL: NCT03139435
Title: A Pilot Study Using Ultrasound for the Detection of Taxane-Induced Peripheral Neuropathy
Brief Title: Ultrasound in Detecting Taxane-Induced Neuropathy in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00043631; NCI-2017-00680 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 97217 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2017-05-01; First posted 2017-05-04 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Peripheral Neuropathy; Stage 0 Breast Cancer; Stage I Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage III Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Carcinoma In Situ; Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (ultrasound) (Experimental): Patients undergo peripheral nerve ultrasound. Patients also undergo skin biopsy.
  Interventions: Procedure: Biopsy; Other: Questionnaire Administration; Diagnostic Test: Ultrasound Tomography

INTERVENTIONS:
Procedure: Biopsy — Undergo skin biopsy
  Other Names: Bx
Other: Questionnaire Administration — Ancillary studies
Diagnostic Test: Ultrasound Tomography — Undergo peripheral nerve ultrasound

SUMMARY:
This pilot clinical trial studies how well ultrasound works in detecting taxane-induced neuropathy in patients with breast cancer. Ultrasound may work better in diagnosing and detecting neuropathy in breast cancer patients treated with the chemotherapy drug called a taxane.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare tibial motor nerve ultrasound cross-sectional area (CSA) between taxane-induced peripheral neuropathy (TIPN) patients and historical data among healthy adults.

SECONDARY OBJECTIVES:

I. To compare sural sensory nerve ultrasound CSA between TIPN patients and historical data among healthy adults.

II. To determine if the above changes in nerve CSA correlate with NCS changes in the same TIPN patients.

III. To determine if the above changes in nerve CSA correlate with changes on a self-reported neuropathy scale (Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20 [QLQ-CIPN20]) in the same TIPN patients.

IV. To determine if the above changes in nerve CSA correlate with intraepidermal nerve fiber (IENF) density changes on skin biopsy in the same TIPN patients.

TERTIARY OBJECTIVES:

I. To assess activated mast cells in skin biopsies in TIPN patients in relation to severity of symptoms and above findings.

II. To assess serum inflammatory markers in TIPN patients in relation to severity of symptoms and above findings.

OUTLINE:

Patients undergo peripheral nerve ultrasound. Patients also undergo skin biopsy.

After completion of study, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer (any stage)
* Previously or currently receiving taxane-based chemotherapy
* Clinical symptoms of peripheral neuropathy noted in medical record and suspected to be secondary to taxane-based therapy
* Ability and willingness to understand and sign an informed consent

Exclusion Criteria:

* Self-reported or documented history of pre-existing peripheral neuropathy prior to initiation of taxane chemotherapy
* Unable to provide history

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Strowd, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Historical control information is a reference group only and were not active participants in this trial.
Units Other Than Participants: nerve samples
Groups:
- Case: Study sample
- Historical Control: Historical Control group - not part of study enrollment
Period: Overall Study
Arm/Group | Case | Historical Control
Started | 20; 20 nerve samples (For those enrolled during the study ('Case'), only one measure per participant is analyzed.) | 60; 120 nerve samples (For the 'Historical Control' arm there are two samples for each participant (one from each arm).)
Completed | 20; 20 nerve samples | 60; 120 nerve samples
Not Completed | 0; 0 nerve samples | 0; 0 nerve samples

BASELINE CHARACTERISTICS:
Units Other Than Participants: nerve samples
Groups:
- Control (From Another Study): These patients were not enrolled as part of this study. This data comes from another study. Each of these n=60 patients had tests done on both left and right arms, which creates the n=120 samples found in the results.
- Total: Total of all reporting groups
Arm/Group | Case | Control (From Another Study) | Total
Number analyzed (Participants) | 20 | 60 | 80
Number analyzed (nerve samples) | 20 | 120 | 140
Age, Continuous [Mean (Full Range); unit: years] | 55.5 [32 to 72] | 45.9 [21 to 80] | 48.3 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 38 | 58
  Male | 0 | 22 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 17 | 55 | 72
  Unknown or Not Reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 0 | 6
  White | 12 | 0 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 60 | 62

OUTCOME MEASURES:

1. Primary Outcome: Tibial Nerve Cross-sectional Area
Description: Will be determined by ultrasound in the tibial nerve. Will be compared to the historical data from healthy patients using two-sample t-test (two-sample t-test selected as primary data from the historical control patients is available and will be used for analysis). Will also compare the nerve cross-sectional area in our study sample to that in the historical diabetic neuropathy patients and historical oxaliplatin neuropathy patients using one-sample t-test. The general linear model will be used to evaluate any factors (e.g., age) that may be associated with the nerve cross-sectional area. Due
Time Frame: Up to 30 days
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: arm
Groups:
- Control: Historical Control
Arm/Group | Case | Control
Number analyzed (Participants) | 20 | 60
Number analyzed (arm) | 20 | 120
mm^2 | 13.0 (3.6) | 14.0 (4.3)

2. Secondary Outcome: Amplitude of Nerve Response - Ankle
Description: Spearman's rank correlation coefficient will be used to examine the associations between nerve cross-sectional area (tibial cross-sectional area) and nerve conduction studies (amplitude of nerve response - ankle).
Time Frame: Up to 30 days
Measure: Number; unit: Spearman correlation coefficient
Units Other Than Participants: arm
Arm/Group | Case
Number analyzed (Participants) | 20
Number analyzed (arm) | 20
Spearman correlation coefficient | 0.15

3. Secondary Outcome: Conduction Velocity of Nerve Response - Tibial
Description: Spearman's rank correlation coefficient will be used to examine the associations between nerve cross-sectional area (tibial cross-sectional area) and nerve conduction studies (conduction velocity of nerve response - tibial).
Time Frame: Up to 30 days
Measure: Number; unit: Spearman correlation coefficient
Units Other Than Participants: arm
Arm/Group | Case
Number analyzed (Participants) | 19
Number analyzed (arm) | 19
Spearman correlation coefficient | 0.15

4. Secondary Outcome: Distal Latency of Nerve Response - Ankle
Description: Spearman's rank correlation coefficient will be used to examine the associations between nerve cross-sectional area (tibial cross-sectional area) and nerve conduction studies (distal latency of nerve response - ankle).
Time Frame: Up to 30 days
Measure: Number; unit: Spearman correlation coefficient
Units Other Than Participants: arm
Arm/Group | Case
Number analyzed (Participants) | 20
Number analyzed (arm) | 20
Spearman correlation coefficient | -0.23

5. Secondary Outcome: Nerve Fiber Density in the Skin
Description: Spearman's rank correlation coefficient will be used to examine the association between nerve cross-sectional area and distal intraepidermal nerve fiber density.
Time Frame: Up to 30 days
Measure: Number; unit: Spearman correlation coefficient
Units Other Than Participants: arm
Arm/Group | Case
Number analyzed (Participants) | 20
Number analyzed (arm) | 20
Spearman correlation coefficient | -0.12

6. Secondary Outcome: Self-reported Neuropathy Score
Description: Will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20. Spearman's rank correlation coefficient will be used to examine the associations between the cross-sectional area and the self-reported neuropathy scale.
Time Frame: Up to 30 days
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | Case
Number analyzed (Participants) | 20
Spearman correlation coefficient | -0.18

7. Secondary Outcome: Sural Nerve Cross-sectional Area
Description: Will be determined by ultrasound of the sural nerve. Spearman's rank correlation coefficient will be used to examine the associations between nerve cross-sectional area and nerve conduction studies. The general linear model will be also used to evaluate the association after adjusting for one or two risk factors (e.g., age). Nerve cross-sectional area will be treated as the dependent variable.
Time Frame: Up to 30 days
Measure: Number; unit: Spearman correlation coefficient
Units Other Than Participants: arm
Arm/Group | Case
Number analyzed (Participants) | 20
Number analyzed (arm) | 20
Spearman correlation coefficient | 0.30

8. Other Pre Specified Outcome: Serum Levels of Inflammatory Molecules
Description: Spearman's rank correlation coefficient will be used to assess the associations between activated mast cells in skin biopsies, serum inflammatory markers, severity of symptoms, and primary outcome and secondary outcomes in taxane-induced peripheral neuropathy patients.
Time Frame: Up to 30 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: The Number of Activated Mast Cells
Description: as for outcome 8
Time Frame: Up to 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 month
Description: Adverse Events were collected during the first treatment cycle. Historical control participants were not a part of this trial and were used as a reference group only. No adverse events were collected from this group.
Arm/Group | Case
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Case (N=20)
Infections and infestations - Other (Infections and infestations) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT03139435/Prot_SAP_001.pdf
  • Informed Consent Form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT03139435/ICF_000.pdf